CLINICAL TRIAL: NCT04845737
Title: Evaluation of the Relationship Between Electrophysiological Findings With Vitamin D Levels and Inflammatory Parameters in Fibromyalgia Patients
Brief Title: Electrophysiological Findings in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, MD, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIBU-FTR-EY-03
Record Dates: First submitted 2021-03-17; First posted 2021-04-15 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia
Keywords: sympathetic skin response; inflammatory parameters; autonomic dysfunction; autonomic nervous system
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: We have two groups.First group is fibromyalgia patient and second group is healty control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia patient group (Other): Sympathetic skin response measurements will be made in patients who meet the diagnosis criteria of fibromyalgia. Vitamin D levels will be measured and hemogram values will be checked in these patients.
  Interventions: Other: sympathetic skin response measurement
- Control Group (Other): The participant in this group will be chosen from healthy volunteers. Sympathetic skin response will be measured of the participants. Vitamin D levels and hemogram values will be recorded.
  Interventions: Other: sympathetic skin response measurement

INTERVENTIONS:
Other: sympathetic skin response measurement — Sympathetic skin response(SSR) was studied with upper and lower extremity hand and foot recording of all participants, and amplitude and latency values will be recorded. SSR measurement will be made at room temperature of 25 ºC, while the patients are resting in the supine position. 6 mm silver disc electrodes will be used as the recording electrode.
  The relationship between the patients' vitamin D levels and inflammatory response markers and their sympathetic skin responses will be investigated by statistical analysis.
  Other Names: measurement of vitamin d levels and hemogram evaluation

SUMMARY:
Fibromyalgia Syndrome (FMS); It is a chronic condition characterized by widespread body pain, sleep disturbance, fatigue, impaired cognitive functions, and anxiety (1). FMS; chronic fatigue syndrome, interstitial cystitis, irritable bowel syndrome, temperomandibular joint dysfunction, myofascial pain, functional dyspepsia, restless leg syndrome and posttraumatic stress disorder are among central sensitization syndromes (2,3).

DETAILED DESCRIPTION:
Etiology and pathogenesis in fibromyalgia have not been fully elucidated. Many mechanisms contribute to the formation of FMS. Many evidence has been found for dysfunction of the central and autonomic nervous system, immune system, cytokines, neurotransmitters and hormones, which are thought to play a role in the disease.

Since increasing systemic inflammation is thought to have a role in the etiopathogenesis of FMS, there are increasing numbers of studies focusing on this aspect of fibromyalgia.

Neutrophil / lymphocyte ratio (NLR) and platelet / lymphocyte ratio (PLR) in peripheral blood are simple markers of systemic inflammatory response.

Another factor thought to have a role in etiopathogenesis is autonomic nervous system dysfunction. It has been found that there is autonomic dysfunction in the sympathetic nervous system in patients with FMS. Sympathetic skin response measurements are frequently used electrophysiological methods to evaluate the functionality of the sympathetic nervous system, which is a component of the autonomic nervous system.

In addition, vitamin D deficiency is common in FMS patients. In a study, inadequate vitamin D levels were found in 45% of fibromyalgia patients.

When a literature review is performed, it is seen that electrophysiological studies are performed to evaluate autonomic dysfunction in patients with fibromyalgia. No studies were found showing the relationship between vitamin D levels and inflammatory parameters in patients with fibromyalgia and electrophysiological findings. In our study, it was aimed to compare the autonomic dysfunction of fibromyalgia patients with healthy volunteers by electrophysiological evaluation and to investigate the relationship between vitamin D levels and inflammatory parameters in fibromyalgia patients and the data obtained from electrophysiological studies. In this way, we aimed to contribute to a better understanding of the physiopathology of fibromyalgia patients with autonomic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old To be diagnosed with FMS according to the criteria of American College of Rheumatology (ACR) 2010 Confirmed diagnosis of FMS according to American College of Rheumatology (ACR) 2016 criteria

Exclusion Criteria:

* Presence of acute infection Diabetes Mellitus B12 deficiency Hypothyroidism Inflammatory-rheumatological disease presence A history of malignancy Major psychiatric disorder Dementia, etc. diseases that may cause loss of cognitive functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Sympathetic Skin Response | 10 minutes
  Sympathetic Skin Response (SSR) measurement will be made at room temperature of 25 ºC, while the patients are resting in the supine position.For upper extremity SSR evaluation, the active (-) electrode will be placed in the palmar area, the reference electrode (+) in the dorsum of the hand, and the ground electrode in the forearm. Similarly, in the lower extremity, the active electrode will be placed on the sole of the foot and the reference electrode will be placed on the back of the foot. The same side median nerve will be stimulated from the second finger, and the SSR obtained from the right upper and lower extremities will be evaluated. The duration of the warning will be adjusted to be 0.1 ms and the intensity of the warning to be 15-20 mA. In order to prevent habituation, warnings will be given at different intervals and with> 30 seconds between warning. A maximum of 5 unilateral stimulation will be applied to each patient.

SECONDARY OUTCOMES:
Visual analogue scale | 45 seconds
  It is used to convert some values that cannot be measured numerically into numerical ones. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by placing a point or pointing on this line.
Fibromyalgia Impact Questionnaire | 60 seconds
  It measures 10 different characteristics: physical function, feeling unwell, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Except for the sense of well-being, lower scores indicate improvement or less affected by the disease. The Fibromyalgia Impact Questionnaire is filled out by the patient. The maximum possible score for each subtitle is 10 points. Thus the total maximum score is 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yakşi, Principal Investigator — Abant İzzet Baysal University Medical Faculty
Locations (1):
- Elif Yakşi, Bolu, Turkey (Türkiye)